CLINICAL TRIAL: NCT01690572
Title: Drug Coated Balloon (DCB) for the Prevention of Constrictive Remodeling and Restenosis in Small Vessel Coronary Disease
Brief Title: Drug Eluting Balloon for Prevention of Constrictive Remodeling
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment was not sufficient.
Sponsor: Prof. Dr. med. Christoph Hehrlein (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Christoph Hehrlein, Professor Dr. med., Herz-Zentrums Bad Krozingen
Organization: Herz-Zentrums Bad Krozingen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEBT
Record Dates: First submitted 2012-09-19; First posted 2012-09-21 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Coronary Disease; Diabetes Mellitus
Keywords: drug eluting balloon; constrictive remodeling
MeSH Terms: conditions — Coronary Disease; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel coated balloon catheter (Active Comparator): Paclitaxel coated balloon catheter "IN.PACT Falcon"
  Interventions: Device: Paclitaxel coated balloon catheter
- uncoated balloon catheter (Active Comparator): uncoated balloon catheter "sprinter legend"
  Interventions: Device: uncoated balloon catheter "sprinter legend"

INTERVENTIONS:
Device: Paclitaxel coated balloon catheter — Dilatation of the target lesion
  Other Names: IN.PACT Falcon
  Arms: Paclitaxel coated balloon catheter
Device: uncoated balloon catheter "sprinter legend" — Dilatation of the target lesion
  Other Names: sprinter legend
  Arms: uncoated balloon catheter

SUMMARY:
Earlier studies indicated that Percutaneous coronary intervention (PCI) may be problematic in diffuse small vessel disease especially of diabetic patients. High restenosis rates after balloon only procedures in small vessels occur due to negative constrictive vessel remodeling if DES (drug eluting stents) are not used and prolonged anti-platelet therapy is not indicated. The main hypothesis of the trial is that in analogy to DCB success in peripheral arterial disease (PAD), cellular toxicity of the drug paclitaxel eluting from a IN.PACT FalconTM DCB will prevent constrictive remodelling of small coronary vessel segments after dilatation. The IN.PACT FalconTM DCB is compared with plain old balloon angioplasty (POBA) using a Sprinter LegendTM balloon in small vessel coronary artery disease. A constrictive remodelling process will be measured by optical coherence tomography (OCT) at 9 months median F/U. This pilot trial is planned to be randomized 1:1 for DCB against POBA therapy.

ELIGIBILITY:
Inclusion Criteria:

* at least one target lesion with a stenosis severity ≥ 50% in one coronary segment with a diameter ≤ 2.5 mm
* age > 18 years
* weight > 45 kg
* patient suitable for balloon dilatation and not suitable for elective implantation of a drug eluting stent
* insulin-dependent or non-insulin-dependent diabetes mellitus
* length of lesion ≥ 15 mm

Exclusion Criteria:

* Life expectancy < 12 months
* In-Stent restenosis
* planned coronary bypass or heart valve OP
* ST elevation myocardial infarction within the last 72 hours
* cardiogenic shock
* renal impairment or liver dysfunction (creatinine > 2.0 mg/dl, AST/ALT > 3x of normal value
* incompliance
* pregnant or breastfeeding women or women who like to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-10; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
MACE-rate | 12 months after initial treatment
  combined end-point: death, myocardial infarction and revascularisation of the target lesion

SECONDARY OUTCOMES:
OCT-measurement | during follow-up, after 9 months
  each symptomatic patient will be examined using optical coherence tomography to detect, if the symptoms are caused by a narrowing at the target lesion

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hehrlein, Prof. Dr., Principal Investigator — Department of Cardiology and Angiology I, Heart Center, Freiburg University
Locations (1):
- Department of Cardiology and Angiology I, Heart Center,, Freiburg im Breisgau, Baden-Wurttemberg, Germany